CLINICAL TRIAL: NCT02648529
Title: Dynamic Regional Brain Maturation in Children With Localization Related Epilepsy
Brief Title: Brain Maturation in Children With Localization Related Epilepsy
Acronym: DYNAMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-700
Record Dates: First submitted 2015-12-02; First posted 2016-01-07 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Benign Childhood Epilepsy With Centro-temporal Spikes (BCECTS); Focal Cryptogenic Epilepsy of Childhood; Cryptogenic Epilepsy of Childhood
Keywords: Benign childhood epilepsy with centro-temporal spikes; rolandic epilepsy; brain development; DTI; functional MRI; structural MRI; idiopathic focal epilepsy; cryptogenic epilepsy of childhood
MeSH Terms: conditions — Epilepsy, Rolandic | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with BCECTS (Experimental): Patients with BCECTS on which MRI, fMRI and neuropsychological assessment will be performed
  Interventions: Procedure: MRI; Procedure: functional MRI (fMRI); Behavioral: neuropsychological assessment
- Healthy volunteers (Other): Healthy volunteers on which MRI, fMRI and neuropsychological assessment will be performed
  Interventions: Procedure: MRI; Procedure: functional MRI (fMRI); Behavioral: neuropsychological assessment

INTERVENTIONS:
Procedure: MRI — Patients are investigated with the following sequences:
  * High-resolution 3D T1-weighted anatomical MRI.
  * DTI with 48 directions (to examine white matter)
Procedure: functional MRI (fMRI) — fMRI investigations will be focused on :
  * language: investigation on possible atypical language networks in children with epilepsy. The fMRI task is a silent verb generation.
  * Social cognition: investigations on social cognition skills
  * Memory :
  * Declarative memory: investigations on the pattern of activations in the brain associated with successful memory formation and changes from childhood to adolescence
  * Working memory: A verbal and a spatial working memory task has been chosen, and is an adaptation of two published cross-sectional studies of working memory from Gabrieli and Sowell groups.
Behavioral: neuropsychological assessment — Patients undergo a repeated annual neuropsychological assessment over the five years of their participation in the project.

SUMMARY:
This project intends to investigate children with idiopathic and cryptogenic localization related epilepsies, using a longitudinal assessment of structural and functional MRI data, in relation to neuropsychological evaluation. The rationale is primarily based on: 1) the frequent observation of selective cognitive dysfunctions in such children, the pathophysiology of which remains largely uncertain; 2) the recent major advances in the MRI investigation of brain maturation showing striking age and region dependant patterns.

The primary hypothesis is that some children with localization related epilepsies suffer from altered maturation in the epileptic brain regions, and that this abnormal maturation affects their cognitive abilities. 100 children with localization related epilepsies and 100 matched controls will be prospectively enrolled during the first two years of the disease (for patients) and benefit from a comprehensive phenotypic and neuropsychological evaluation once a year for 5 years. The brain maturation of these children will be longitudinally assessed using structural and functional MRI, and correlated with neuropsychological data. Investigators hope to demonstrate that children with localization related epilepsies and cognitive dysfunctions suffer from an abnormal brain maturation in regions underlying the epileptic activity and the altered cognitive processes. The finding could partly bridge the gap between these two abnormalities and help better understand their interaction and respective dynamic. Once validated, the study of regional brain maturation in children with epilepsy might be further used as a reliable surrogate marker or predictor of associated cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* motivation to participate in the study for 5 years
* for patients - one of the following diagnostics - BCECTS (benign childhood epilepsy with centro-temporal spikes), focal cryptogenic epilepsy of childhood, Panayiotopoulos syndrome, diagnosis established according to the current diagnostic criteria (ILAE, 1989)
* for patients - no anti-epileptic drug for 24 months
* normal MRI if available before inclusion
* signed consent by on of the parents

Exclusion Criteria:

* associated neurological and psychiatric diseases
* other epileptic syndromes
* other chronic severe disease
* contra-indication for performing an MRI examination
* claustrophobia

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2008-09; Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Rate of grey/white matter volume | At 5 years
  The aim is to evaluate structural brain maturation. All subjects will benefit from a 3D-T1 1,5 Tesla MRI and 48-directions Diffusion Tensor Imaging (DTI). We will calculate parametric maps of individual regional changes of grey/white matter fractions over time. This study aims to detect a significant difference in the rate of grey/white matter volume change over the epileptic region. We will further correlate a number of neuropsychological and clinical variables with the parametric maps of brain maturation. There will be annual measures up to 5 years after inclusion.

SECONDARY OUTCOMES:
Changes in fMRI activation of language areas in brain during cognitive tasks | At 5 years
  The aim is to evaluate functional brain maturation of language. All subjects will benefit from the functional MRI (fMRI) evaluation of the cognitive tasks. Changes in fMRI activation over time will be studied at the group level, taking into account all potentially relevant variables. This outcomme will be assessed at year 1, 3 and 5 after inclusion.
Changes in fMRI activation of social cognition areas in brain during cognitive tasks | At 5 years
  The aim is to evaluate functional Brain Maturation of social cognition. All subjects will benefit from the functional MRI (fMRI) evaluation of the cognitive tasks. Changes in fMRI activation over time will be studied at the group level, taking into account all potentially relevant variables. This outcomme will be assessed at year 1, 3 and 5 after inclusion.
Changes in fMRI activation of Working memory areas in brain during cognitive tasks | At 5 years
  The aim is to evaluate Functional Brain Maturation of Working memory. All subjects will benefit from the functional MRI (fMRI) evaluation of the cognitive tasks. Changes in fMRI activation over time will be studied at the group level, taking into account all potentially relevant variables. This outcomme will be assessed at year 1, 3 and 5 after inclusion.
Changes in fMRI activation of declarative memory areas in brain during cognitive tasks | At 5 years
  The aim is to evaluate Functional Brain Maturation of declarative memory. All subjects will benefit from the functional MRI (fMRI) evaluation of the cognitive tasks. Changes in fMRI activation over time will be studied at the group level, taking into account all potentially relevant variables. This outcomme will be assessed at year 1, 3 and 5 after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain RHEIMS, Principal Investigator — Service d'épileptologie fonctionnelle, Hôpital Pierre Wertheimer, Hospices Civils de Lyon
Locations (1):
- Hôpital Femme-Mère-Enfant, 59 Boulevard Pinel, Bron, France